CLINICAL TRIAL: NCT00617344
Title: Immunogenicity and Safety of Three Tetravalent Formulations of Dengue Vaccine Candidates in Healthy Adults Aged 18 to 45 Years in the US
Brief Title: Immunogenicity and Safety of Three Formulations of Dengue Vaccines in Healthy Adults Aged 18 to 45 Years in the US
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CYD12
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Dengue Virus
Keywords: Dengue fever; Dengue hemorrhagic fever; Dengue virus
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CYD Dengue Vaccine 5555 Formulation (Experimental): Participants received 3 doses of CYD dengue vaccine (5555 formulation); one each at 0 (vaccination 1), 6 (vaccination 2), and 12 (vaccination 3) months.
  Interventions: Biological: Tetravalent CYD Dengue Vaccine , 5555 formulation
- CYD Dengue Vaccine 5553 Formulation (Experimental): Participants received 3 doses of CYD dengue vaccine (5553 formulation); one each at 0 (vaccination 1), 6 (vaccination 2), and 12 (vaccination 3) months.
  Interventions: Biological: Tetravalent CYD Dengue Vaccine , 5553 formulation
- CYD Dengue Vaccine 4444 Formulation (Experimental): Participants received 3 doses of CYD dengue vaccine (4444 formulation); one each at 0 (vaccination 1), 6 (vaccination 2), and 12 (vaccination 3) months.
  Interventions: Biological: Tetravalent CYD Dengue Vaccine, 4444 formulation

INTERVENTIONS:
Biological: Tetravalent CYD Dengue Vaccine , 5555 formulation — A 0.5 mL dose, Subcutaneous at 0, 6, and 12 months, respectively.
  Arms: CYD Dengue Vaccine 5555 Formulation
Biological: Tetravalent CYD Dengue Vaccine , 5553 formulation — A 0.5 mL dose, Subcutaneous at 0, 6, and 12 months, respectively
  Arms: CYD Dengue Vaccine 5553 Formulation
Biological: Tetravalent CYD Dengue Vaccine, 4444 formulation — A 0.5 mL dose, Subcutaneous at 0, 6, and 12 months, respectively
  Arms: CYD Dengue Vaccine 4444 Formulation

SUMMARY:
This study used 3 different formulations of tetravalent CYD dengue vaccine.

The primary objective of the study was to evaluate the neutralizing antibody response after 2 doses of two different formulations of tetravalent dengue vaccine administered at Month 0 and Month 6.

The secondary objectives were:

* To evaluate the safety of the 3 formulations of tetravalent CYD dengue vaccine.
* To describe the neutralizing antibody responses to each of the 3 vaccine formulations.
* To describe vaccine viremia after the first and second dose of each of the 3 vaccine formulations in a subset of participants.

DETAILED DESCRIPTION:
All participants provided blood samples for immunogenicity assessments, while vaccine viremia was assessed in a subset of participants in each group.

Safety was assessed in all participants as follows: solicited adverse event (AE) prelisted in the diary card were collected for 7 days after vaccination for solicited injection site reactions and 14 days for solicited systemic reactions , unsolicited AEs were collected for 28 days after vaccination, and serious adverse event (SAE) information collected throughout the study up to 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history, clinical examination, and biological safety parameters.
* Aged 18 to 45 years on the day of inclusion.
* Provision of informed consent signed by the participant or another legally acceptable representative.
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination, and until at least 4 weeks after the last study vaccination.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* For a woman of child-bearing potential, known or suspected pregnancy or positive serum/urine pregnancy test.
* Breast-feeding woman.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term (at least 2 weeks within the previous 3 months) systemic corticosteroids therapy (at a dose of at least 10 mg). Topical steroids were allowed.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator.
* Current or past alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following each of the trial vaccinations.
* Human Immunodeficiency Virus (HIV), hepatitis B surface antigen, or hepatitis C virus seropositivity in blood sample taken at Screening.
* Participant deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Clinically significant laboratory test abnormalities (as determined by the investigator) in blood sample taken at Screening.
* Previous residence in, travel or planned travel of more than 2 weeks during the study period to areas with high dengue infection endemicity.
* Reported history of flavivirus infection as reported by the participant.
* Previous vaccination against flavivirus diseases (including Japanese encephalitis, tick-borne encephalitis, and yellow fever).
* Flavivirus vaccination planned during the trial period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2008-04-17 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (5):
- United States (5):
  - Investigational Site 004, Hoover, Alabama
  - Investigational Site 002, San Diego, California
  - Investigational Site 005, Vallejo, California
  - Investigational Site 001, New Orleans, Louisiana
  - Investigational Site 003, Springfield, Missouri

REFERENCES:
- [Result] Dayan GH, Thakur M, Boaz M, Johnson C. Safety and immunogenicity of three tetravalent dengue vaccine formulations in healthy adults in the USA. Vaccine. 2013 Oct 17;31(44):5047-54. doi: 10.1016/j.vaccine.2013.08.088. Epub 2013 Sep 7. PMID 24021313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 17 April 2008 to 04 June 2008 at 5 sites in the United States.
Pre-assignment Details: A total of 309 participants were screened in the study, out of which 260 participants were enrolled and vaccinated in the study. Screen failures were mainly due to inclusion criteria not met or exclusion criteria met.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Started | 104 | 103 | 53
Received Vaccination 1 | 104 | 103 | 53
Received Vaccination 2 | 86 | 85 | 46
Received Vaccination 3 | 79 | 81 | 45
Completed | 79 | 81 | 45
Not Completed | 25 | 22 | 8
Not completed — Serious adverse event | 1 | 0 | 0
Not completed — Other Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 10 | 8 | 5
Not completed — Lost to Follow-up | 5 | 4 | 1
Not completed — Withdrawal by Subject | 8 | 9 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all the participants enrolled in the trial who received at least 1 injection of CYD Dengue Vaccine and had any valid immunogenicity result.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation | Total
Number analyzed (Participants) | 101 | 101 | 53 | 255
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.6 (8.78) | 32.1 (8.57) | 32.4 (8.04) | 32.4 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 32 | 152
  Male | 40 | 42 | 21 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers of >= 10 1/Dilution (1/Dil) Against Each Dengue Virus Serotype Strain: CYD Vaccine 5555 and 5553 Formulation
Description: Percentage of participants with antibody titers >= 10 (1/dil) against each serotypes (1, 2, 3 and 4) of the dengue virus strains was assessed by dengue plaque reduction neutralization test (PRNT).
Time Frame: Pre-injection 1 (Day 0), 30 days post-injection 2 (Month 7)
Population: Analysis was performed on Full Analysis Set (FAS). Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation
Number analyzed (Participants) | 101 | 101
percentage of participants
  Dengue Virus Serotype 1: Day 0 | 1.0 | 3.0
  Dengue Virus Serotype 1:30 days post injection-2: number analyzed (Participants) | 81 | 84
  Dengue Virus Serotype 1:30 days post injection-2 | 65.4 | 81.0
  Dengue Virus Serotype 2: Day 0 | 1.0 | 3.0
  Dengue Virus Serotype 2:30 days post-injection 2: number analyzed (Participants) | 81 | 84
  Dengue Virus Serotype 2:30 days post-injection 2 | 80.2 | 83.3
  Dengue Virus Serotype 3: Day 0 | 15.8 | 14.9
  Dengue Virus Serotype 3:30 days post-injection 2: number analyzed (Participants) | 78 | 84
  Dengue Virus Serotype 3:30 days post-injection 2 | 87.2 | 92.9
  Dengue Virus Serotype 4: Day 0 | 3.0 | 6.9
  Dengue Virus Serotype 4:30 days post-injection 2: number analyzed (Participants) | 78 | 84
  Dengue Virus Serotype 4:30 days post-injection 2 | 89.7 | 58.3
Statistical Analysis 1: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 1: Pre-injection 1 (Day 0); Test type: Other — The associated 95% confidence intervals (CIs) for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -2.0, 95% CI 2-sided [-7.44 to 2.84]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 1: 30 days post-injection 2; Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -15.5, 95% CI 2-sided [-28.4 to -2.00]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 2: Pre-injection 1 (Day 0); Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -2.0, 95% CI 2-sided [-7.44 to 2.84]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 2: 30 days post-injection 2; Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -3.1, 95% CI 2-sided [-15.0 to 8.75]
Statistical Analysis 5: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 3: Pre-injection 1 (Day 0); Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = 1.0, 95% CI 2-sided [-9.09 to 11.1]
Statistical Analysis 6: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 3: 30 days post-injection 2; Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -5.7, 95% CI 2-sided [-15.6 to 3.81]
Statistical Analysis 7: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 4: Pre-injection 1 (Day 0); Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = -4.0, 95% CI 2-sided [-10.9 to 2.49]
Statistical Analysis 8: Comparison: CYD Dengue Vaccine 5555 Formulation vs CYD Dengue Vaccine 5553 Formulation; Dengue Virus Serotype 4: 30 days post-injection 2; Test type: Other — The associated 95% CIs for the point estimates and the differences were calculated using normal approximation; Difference in Percentage = 31.4, 95% CI 2-sided [18.2 to 43.2]

2. Secondary Outcome: Percentage of Participants With Antibody Titers of >=10 1/Dil Against Each Dengue Virus Serotype Strain
Description: Percentage of participants with antibody titers >= 10 1/dil against each serotypes (1, 2, 3 and 4) of the dengue virus strains was assessed by PRNT.
Time Frame: Pre-injection 1 (Day 0), 30 days post-injection 1(Month 1), injection 2 (Month 7) and injection 3 (Month 13)
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 101 | 101 | 53
percentage of participants
  Dengue Virus Serotype 1: Day 0 | 1.0 | 3.0 | 3.8
  Dengue Virus Serotype 1:30 days post-injection 1 | 33.7 | 50.5 | 26.4
  Dengue Virus Serotype 1:30 days post-injection 2: number analyzed (Participants) | 81 | 84 | 46
  Dengue Virus Serotype 1:30 days post-injection 2 | 65.4 | 81.0 | 58.7
  Dengue Virus Serotype 1:30 days post-injection 3: number analyzed (Participants) | 69 | 81 | 45
  Dengue Virus Serotype 1:30 days post-injection 3 | 71.0 | 84.0 | 64.4
  Dengue Virus Serotype 2: Day 0 | 1.0 | 3.0 | 1.9
  Dengue Virus Serotype 2:30 days post-injection 1 | 46.5 | 64.4 | 34.0
  Dengue Virus Serotype 2:30 days post-injection 2: number analyzed (Participants) | 81 | 84 | 46
  Dengue Virus Serotype 2:30 days post-injection 2 | 80.2 | 83.3 | 58.7
  Dengue Virus Serotype 2:30 days post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  Dengue Virus Serotype 2:30 days post-injection 3 | 84.3 | 88.9 | 77.8
  Dengue Virus Serotype 3: Day 0 | 15.8 | 14.9 | 13.2
  Dengue Virus Serotype 3:30 days post-injection 1 | 79.2 | 80.2 | 60.4
  Dengue Virus Serotype 3:30 days post-injection 2: number analyzed (Participants) | 78 | 84 | 46
  Dengue Virus Serotype 3:30 days post-injection 2 | 87.2 | 92.9 | 78.3
  Dengue Virus Serotype 3:30 days post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  Dengue Virus Serotype 3:30 days post-injection 3 | 88.6 | 98.8 | 82.2
  Dengue Virus Serotype 4: Day 0 | 3.0 | 6.9 | 5.7
  Dengue Virus Serotype 4:30 days post-injection 1 | 84.2 | 37.6 | 94.3
  Dengue Virus Serotype 4:30 days post-injection 2: number analyzed (Participants) | 78 | 84 | 46
  Dengue Virus Serotype 4:30 days post-injection 2 | 89.7 | 58.3 | 89.1
  Dengue Virus Serotype 4:30 days post-injection 3: number analyzed (Participants) | 69 | 81 | 45
  Dengue Virus Serotype 4:30 days post-injection 3 | 94.2 | 69.1 | 93.3

3. Secondary Outcome: Percentage of Participants With Antibody Titers >=10 1/Dil Against At Least Any 1, 2, 3 or All 4 Dengue Virus Serotypes
Description: Percentage of participants with antibody titers >= 10 1/dil against each serotypes (1, 2, 3 and 4) of the dengue virus strains was assessed by PRNT. In this outcome measure, participants with antibody titers >= 10 1/dil against any 1 of the 4 serotypes or any 2 of the 4 serotypes or any 3 of the 4 serotypes or with all 4 serotypes were reported.
Time Frame: Pre-injection 1 (Day 0), 30 days post-injection 1(Month 1), injection 2 (Month 7) and injection 3 (Month 13)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 101 | 101 | 53
percentage of participants
  At least 1 positive serotype: Day 0 | 16.8 | 20.8 | 17.0
  At least 1 positive serotype: Post-injection 1 | 96.0 | 93.1 | 98.1
  At least 1 positive serotype: Post-injection 2: number analyzed (Participants) | 82 | 84 | 46
  At least 1 positive serotype: Post-injection 2 | 97.6 | 97.6 | 97.8
  At least 1 positive serotype: Post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  At least 1 positive serotype: Post-injection 3 | 100.0 | 100.0 | 100.0
  At least 2 positive serotype: Day 0 | 3.0 | 3.0 | 3.8
  At least 2 positive serotype: Post-injection 1 | 80.2 | 74.3 | 64.2
  At least 2 positive serotype: Post-injection 2: number analyzed (Participants) | 82 | 84 | 46
  At least 2 positive serotype: Post-injection 2 | 90.2 | 90.5 | 82.6
  At least 2 positive serotype: Post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  At least 2 positive serotype: Post-injection 3 | 90.0 | 95.1 | 91.1
  At least 3 positive serotype: Day 0 | 1.0 | 2.0 | 1.9
  At least 3 positive serotype: Post-injection 1 | 50.5 | 45.5 | 41.5
  At least 3 positive serotype: Post-injection 2: number analyzed (Participants) | 82 | 84 | 46
  At least 3 positive serotype: Post-injection 2 | 72.0 | 79.8 | 63.0
  At least 3 positive serotype: Post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  At least 3 positive serotype: Post-injection 3 | 82.9 | 86.4 | 73.3
  All 4 positive serotype: Day 0 | 0.0 | 2.0 | 1.9
  All 4 positive serotype: Post-injection 1 | 16.8 | 19.8 | 11.3
  All 4 positive serotype: Post-injection 2: number analyzed (Participants) | 82 | 84 | 46
  All 4 positive serotype: Post-injection 2 | 52.4 | 47.6 | 41.3
  All 4 positive serotype: Post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  All 4 positive serotype: Post-injection 3 | 62.9 | 59.3 | 53.3

4. Secondary Outcome: Geometric Means of Titers of Antibodies Against Each Dengue Virus Serotype Strain
Description: Geometric mean titers against each dengue virus serotype (1, 2, 3 and 4) strain was measured by PRNT.
Time Frame: Pre-injection 1 (Day 0), 30 days post-injection 1(Month 1), injection 2 (Month 7) and injection 3 (Month 13)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 101 | 101 | 53
Titers (1/dil)
  Dengue Virus Serotype 1: Day 0 | 5.04 [4.96 to 5.13] | 5.57 [4.88 to 6.36] | 5.23 [4.90 to 5.58]
  Dengue Virus Serotype 1:30 days post-injection 1 | 9.97 [8.11 to 12.3] | 20.3 [14.6 to 28.2] | 9.29 [6.51 to 13.3]
  Dengue Virus Serotype 1:30 days post-injection 2: number analyzed (Participants) | 81 | 84 | 46
  Dengue Virus Serotype 1:30 days post-injection 2 | 24.1 [18.1 to 32.1] | 45.4 [33.7 to 61.2] | 19.2 [12.4 to 29.8]
  Dengue Virus Serotype 1:30 days post-injection 3: number analyzed (Participants) | 69 | 81 | 45
  Dengue Virus Serotype 1:30 days post-injection 3 | 24.4 [18.5 to 32.1] | 57.1 [42.2 to 77.3] | 24.2 [15.8 to 37.2]
  Dengue Virus Serotype 2: Day 0 | 5.13 [4.87 to 5.40] | 5.53 [4.93 to 6.20] | 5.43 [4.60 to 6.42]
  Dengue Virus Serotype 2:30 days post-injection 1 | 16.7 [12.3 to 22.6] | 39.9 [27.9 to 57.3] | 13.1 [8.60 to 20.0]
  Dengue Virus Serotype 2:30 days post-injection 2: number analyzed (Participants) | 81 | 84 | 46
  Dengue Virus Serotype 2:30 days post-injection 2 | 47.5 [33.4 to 67.4] | 91.9 [60.7 to 139] | 31.8 [18.6 to 54.3]
  Dengue Virus Serotype 2:30 days post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  Dengue Virus Serotype 2:30 days post-injection 3 | 54.8 [38.7 to 77.7] | 102 [72.7 to 143] | 46.5 [29.1 to 74.2]
  Dengue Virus Serotype 3: Day 0 | 6.60 [5.78 to 7.53] | 6.85 [5.82 to 8.05] | 6.25 [5.30 to 7.37]
  Dengue Virus Serotype 3:30 days post-injection 1 | 45.5 [34.0 to 60.9] | 109 [70.9 to 169] | 23.3 [15.2 to 35.5]
  Dengue Virus Serotype 3:30 days post-injection 2: number analyzed (Participants) | 78 | 84 | 46
  Dengue Virus Serotype 3:30 days post-injection 2 | 64.5 [48.3 to 86.1] | 117 [86.9 to 159] | 40.4 [26.3 to 62.1]
  Dengue Virus Serotype 3:30 days post-injection 3: number analyzed (Participants) | 70 | 81 | 45
  Dengue Virus Serotype 3:30 days post-injection 3 | 63.5 [46.9 to 85.9] | 114 [90.9 to 143] | 43.1 [29.1 to 63.8]
  Dengue Virus Serotype 4: Day 0 | 5.26 [4.96 to 5.59] | 5.57 [5.12 to 6.06] | 5.43 [4.92 to 5.99]
  Dengue Virus Serotype 4:30 days post-injection 1 | 438 [273 to 704] | 12.1 [9.26 to 15.9] | 643 [370 to 1117]
  Dengue Virus Serotype 4:30 days post-injection 2: number analyzed (Participants) | 78 | 84 | 46
  Dengue Virus Serotype 4:30 days post-injection 2 | 150 [104 to 215] | 18.3 [13.6 to 24.7] | 164 [99.4 to 272]
  Dengue Virus Serotype 4:30 days post-injection 3: number analyzed (Participants) | 69 | 81 | 45
  Dengue Virus Serotype 4:30 days post-injection 3 | 133 [98.6 to 179] | 25.9 [18.7 to 36.0] | 134 [86.3 to 207]

5. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions After Any Vaccination
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Pain: Grade 1: Easily tolerated, Grade 2: Sufficiently discomforting to interfere with normal behavior or activities, Grade 3: Incapacitating, unable to perform usual activities. Erythema:- Grade 1: <2.5 cm, Grade 2: >=2.5 to <5 cm, Grade 3: >=5 cm. Swelling:- Grade 1: <2.5 cm, Grade 2: >=2.5 to <5 cm, Grade 3: >=5 cm.
Time Frame: 7 days after any injection 1, 2 or 3
Population: Analysis was performed on Safety Analysis Set which included all participants included in the trial who had received at least 1 dose of study vaccine and had any available safety data. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 101 | 101 | 53
Participants
  Pain: number analyzed (Participants) | 100 | 101 | 52
  Pain | 50 | 42 | 15
  Pain: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Pain: Grade 1 | 46 | 35 | 15
  Pain: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Pain: Grade 2 | 3 | 7 | 0
  Pain: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Pain: Grade 3 | 1 | 0 | 0
  Erythema: number analyzed (Participants) | 100 | 101 | 52
  Erythema | 26 | 27 | 8
  Erythema: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Erythema: Grade 1 | 18 | 19 | 8
  Erythema: Grade 2: number analyzed (Participants) | 100 | 101 | 53
  Erythema: Grade 2 | 7 | 7 | 0
  Erythema: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Erythema: Grade 3 | 1 | 1 | 0
  Swelling: number analyzed (Participants) | 100 | 101 | 52
  Swelling | 19 | 14 | 3
  Swelling: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Swelling: Grade 1 | 15 | 12 | 3
  Swelling: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Swelling: Grade 2 | 3 | 2 | 0
  Swelling: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Swelling: Grade 3 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Solicited Systemic Reactions After Any Vaccination
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Fever: - Grade1: >=37.5°C to <=38.0°C (>=99.5°F to <=100.4°F), Grade 2: >38.0°C to <=39.0°C (>100.4°F to <= 102.2°F), Grade 3: >39.0°C (>102.2°F). Headache, malaise, myalgia and asthenia: Grade 1: noticeable but does not interfere with daily activities, Grade 2: interferes with daily activities, Grade 3: prevents daily activities.
Time Frame: 14 days after any injection 1, 2 or 3
Population: Analysis was performed on safety analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 101 | 101 | 53
Participants
  Fever | 14 | 20 | 6
  Fever: Grade 1 | 11 | 18 | 3
  Fever: Grade 2 | 2 | 2 | 3
  Fever: Grade 3 | 1 | 0 | 0
  Headache: number analyzed (Participants) | 100 | 101 | 52
  Headache | 58 | 59 | 28
  Headache: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Headache: Grade 1 | 28 | 38 | 16
  Headache: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Headache: Grade 2 | 24 | 18 | 9
  Headache: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Headache: Grade 3 | 6 | 3 | 3
  Malaise: number analyzed (Participants) | 100 | 101 | 52
  Malaise | 39 | 43 | 14
  Malaise: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Malaise: Grade 1 | 16 | 26 | 9
  Malaise: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Malaise: Grade 2 | 19 | 12 | 5
  Malaise: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Malaise: Grade 3 | 4 | 5 | 0
  Myalgia: number analyzed (Participants) | 100 | 101 | 52
  Myalgia | 43 | 49 | 18
  Myalgia: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Myalgia: Grade 1 | 29 | 30 | 10
  Myalgia: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Myalgia: Grade 2 | 10 | 17 | 7
  Myalgia: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Myalgia: Grade 3 | 4 | 2 | 1
  Asthenia: number analyzed (Participants) | 100 | 101 | 52
  Asthenia | 29 | 32 | 12
  Asthenia: Grade 1: number analyzed (Participants) | 100 | 101 | 52
  Asthenia: Grade 1 | 18 | 17 | 9
  Asthenia: Grade 2: number analyzed (Participants) | 100 | 101 | 52
  Asthenia: Grade 2 | 8 | 14 | 3
  Asthenia: Grade 3: number analyzed (Participants) | 100 | 101 | 52
  Asthenia: Grade 3 | 3 | 1 | 0

7. Secondary Outcome: Number of Participants With Vaccine Viremia
Description: Vaccine viremia (level of vaccine virus in blood samples taken from participants) was measured by an assay yellow fever reverse transcriptase polymerase chain reaction which allowed the detection of vaccine viremia of any serotype (1, 2, 3 and 4).
Time Frame: 7 days post-injection 1 and 2, 14 days post-injection 1 and 2
Population: Analysis was performed on Viremia Analysis Set which included all participants who received study vaccination and provided at least one blood sample for which vaccine viremia laboratory results were available. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Vaccine viremia 7 days post-injection 1: number analyzed (Participants) | 26 | 25 | 26
  Vaccine viremia 7 days post-injection 1 | 0 | 0 | 0
  Vaccine viremia 14 days post-injection 1: number analyzed (Participants) | 25 | 26 | 26
  Vaccine viremia 14 days post-injection 1 | 0 | 0 | 0
  Vaccine viremia 7 days post-injection 2: number analyzed (Participants) | 25 | 20 | 21
  Vaccine viremia 7 days post-injection 2 | 0 | 0 | 0
  Vaccine viremia 14 days post-injection 2: number analyzed (Participants) | 25 | 20 | 22
  Vaccine viremia 14 days post-injection 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 28 days after each dose of CYD dengue vaccine or Placebo. Solicited Reaction (SR) data were collected within 7 and 14 days after each vaccination. Serious adverse event (SAE) data were collected throughout the study, up to 6 months after last vaccination (up to 18 months).
Description: Analysis was performed on Safety Analysis Set.
Arm/Group | CYD Dengue Vaccine 5555 Formulation | CYD Dengue Vaccine 5553 Formulation | CYD Dengue Vaccine 4444 Formulation
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/101 | 3/101 | 1/53
Other Adverse Events (participants affected / at risk) | 78/101 | 82/101 | 39/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine 5555 Formulation (N=101) | CYD Dengue Vaccine 5553 Formulation (N=101) | CYD Dengue Vaccine 4444 Formulation (N=53)
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Optic Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine 5555 Formulation (N=101) | CYD Dengue Vaccine 5553 Formulation (N=101) | CYD Dengue Vaccine 4444 Formulation (N=53)
Asthenia (General disorders) | 29 (38) | 32 (41) | 12 (14)
Injection Site Erythema (General disorders) | 26 (36) | 27 (34) | 8 (11)
Injection Site Pain (General disorders) | 50 (73) | 42 (64) | 16 (21)
Injection Site Swelling (General disorders) | 19 (23) | 14 (14) | 3 (4)
Malaise (General disorders) | 39 (63) | 43 (57) | 14 (17)
Pyrexia (General disorders) | 14 (17) | 21 (25) | 6 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 7 (7) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 43 (68) | 50 (72) | 18 (21)
Headache (Nervous system disorders) | 59 (104) | 60 (94) | 28 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.